CLINICAL TRIAL: NCT04065932
Title: A Study to Determine the Pharmacokinetic Profile of BMS-986165 Administered as Various Solid Dispersion Tablet Formulations in Healthy Subjects
Brief Title: A Study to Determine the Pharmacokinetic Profile of BMS-986165 Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM011-020
Record Dates: First submitted 2019-08-21; First posted 2019-08-22 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Lupus
MeSH Terms: interventions — deucravacitinib; Famotidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- BMS-985165-01 prototype formulation 1 (Experimental)
  Interventions: Drug: BMS-986165-01
- BMS-986165 Tablet (Experimental)
  Interventions: Drug: BMS-986165 Tablet
- BMS-985165-01 prototype formulation 2 (Experimental)
  Interventions: Drug: BMS-986165-01
- BMS-985165-01 prototype formulation 3 (Experimental)
  Interventions: Drug: BMS-986165-01
- BMS-985165-01 prototype formulation 3 or 4 (Experimental)
  Interventions: Drug: BMS-986165-01; Drug: Famotidine
- BMS-985165-01 prototype formulation 3, 4 or 5 (Experimental)
  Interventions: Drug: BMS-986165-01; Drug: Famotidine

INTERVENTIONS:
Drug: BMS-986165-01 — Participants will receive BMS- 986165 -01 in prototype formulation
  Arms: BMS-985165-01 prototype formulation 1; BMS-985165-01 prototype formulation 2; BMS-985165-01 prototype formulation 3; BMS-985165-01 prototype formulation 3 or 4; BMS-985165-01 prototype formulation 3, 4 or 5
Drug: BMS-986165 Tablet — Participants will receive BMS-986165 in tablet form.
  Arms: BMS-986165 Tablet
Drug: Famotidine — Participants will receive a previously dosed BMS-985165-01 Prototype Tablet at the same dose level following administration of famotidine
  Arms: BMS-985165-01 prototype formulation 3 or 4; BMS-985165-01 prototype formulation 3, 4 or 5

SUMMARY:
A Study to Determine the Drug Level Profile of Different formulations of BMS-986165 Tablets

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patients must be willing and able to complete all study-specific procedures and visits
* Healthy patients, as determined by no clinically significant deviation from normal in medical history, physical examination, electrocardiogram, and clinical laboratory determinations
* Body mass index (BMI) of 18 to 32 kg/m2, inclusive, at screening
* Normal renal function at screening

Exclusion Criteria:

* History or presence of chronic bacterial, viral infection, or autoimmune disorder
* Active TB requiring treatment or documented latent TB within the previous 3 years
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect absorption
* WOCBP (women of childbearing potential) must have negative serum or urine pregnancy test.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2019-12-08 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) for BMS-986165 | Day 1 of treatment
Area under the serum concentration-time curve from time zero to time of last quantifiable concentration- AUC(0-T) for BMS- 986165 | Day 1 of treatment
Area under the plasma concentration-time curve from time zero extrapolated to infinite time- AUC(INF) for BMS-986165 | Day 1 of treatment

SECONDARY OUTCOMES:
Time to maximum observed plasma concentration-(Tmax) for BMS -986165 | Day 1 of treatment
Apparent plasma elimination half-life- (T-HALF) for BMS-986165 | Day 1 of treatment
Area under the concentration-time curve from time zero to 24 hours post- (AUC 0-24) for BMS-986165 | Day 1 of treatment
Apparent clearance -(CL/F) for BMS-986165 | Day 1 of treatment
Concentration observed at 24 hours-(C24) for BMS-986165 | Day 1 of treatment
Concentration observed at 12 hours-(C12) for BMS-986165 | Day 1 of treatment
Incidence of non-serious adverse events(AE's) leading to discontinuation of study therapy. | Approximately 16 weeks
Incidence of serious adverse events (SAE) leading to discontinuation of study therapy. | Approximately 16 weeks.
Incidence of adverse events (AEs) leading to discontinuation of study therapy. | Approximately 16 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Quotient Sciences, Nottingham, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm